CLINICAL TRIAL: NCT05961501
Title: The Evaluation of the Effectiveness of Cannabidiol (CBD) and Cannabinol (CBN) Oral Solutions in the Treatment of Facial Pain and Headache of Muscular Origin
Brief Title: The Effectiveness of CBD and CBN in the Treatment of Facial Pain and Headache of Muscular Origin
Status: Enrolling by invitation | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Wroclaw Medical University (Other)
Responsible Party: Principal Investigator, Joanna Smardz, Investigator, Wroclaw Medical University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: WMU1/2023
Record Dates: First submitted 2023-05-25; First posted 2023-07-27 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-07

CONDITIONS: Myalgia; Muscle Pain; Orofacial Pain; Headache, Tension; Headaches Muscular; Headache
Keywords: cannabidiol; cannabinol
MeSH Terms: conditions — Myalgia; Facial Pain; Tension-Type Headache; Headache | interventions — Cannabinol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Study Group (Experimental): Participants with facial pain and headache of muscular origin which last for more than 3 months. Each of the participants in this group will receive the aqueous solution of CBD and CBN to drink in home every day for 60 days in a specific dose determined by the attending physician
  Interventions: Drug: An aqueous solution containing CBD and CBN
- Control group (Placebo Comparator): Participants with facial pain and headache of muscular origin which last for more than 3 months. Each of the participants in this group will receive the placebo to drink in home every day for 60 days in a specific dose determined by the attending physician
  Interventions: Other: The aqueous solution of placebo

INTERVENTIONS:
Drug: An aqueous solution containing CBD and CBN — An aqueous solution containing CBD and CBN, to drink at home in the dose determined by the attending physician
  Arms: Study Group
Other: The aqueous solution of placebo — An aqueous solution of placebo, to drink at home in the dose determined by the attending physician
  Arms: Control group

SUMMARY:
The aim of the study is to evaluate the effectiveness of an aqueous solution containing CBD and CBN in the management of Facial Pain and Headache of Muscular Origin. A randomized (block randomization), double-blind, two-arm controlled trial will involve 42 adult patients diagnosed with Facial Pain and Headache of Muscular Origin which is lasting more than 3 months on the basis of clinical examination. Qualified study participants will be randomly assigned to two groups. The studied group will receive tan aqueous solution containing CBD and CBN, to drink at home in the dose determined by the attending physician, while the control group will receive an aqueous solution of placebo, to drink at home in the dose determined by the attending physician during this time. Each subject will be tested on the qualification day (D0), on 20 days after D0 (D20), and then 40 (D40) and 60 (D60) days after the qualification day using electromyography (EMG), pressure pain threshold test (PPT), clinical examination and surveys.

DETAILED DESCRIPTION:
Background: Orofacial pain is a common occurrence. According to available scientific research, it occurs in up to 16 to 25% of the human population. In its chronic form, orofacial pain can lead to reduced sleep quality, reduced life satisfaction, and psychoemotional disorders, including depressive disorders. A popular tendency among patients suffering from chronic orofacial pain is the abuse of non-steroidal anti-inflammatory drugs, which in most cases show low, short-term and disproportionate to side effects effectiveness. There are scientific reports suggesting that substances such as cannabidiol (CBD) and cannabinol (CBN) may be effective in the treatment of chronic nociceptive and neuropathic pain. However, studies on the effectiveness of these substances in alleviating muscular orofacial pain are clearly lacking

Aim: The aim of the study is to evaluate the effectiveness of an aqueous solution containing CBD and CBN in the management of Facial Pain and Headache of Muscular Origin

Material and methods: A randomized (block randomization), double-blind, two-arm controlled trial will involve 42 adult patients diagnosed with Facial Pain and Headache of Muscular Origin which is lasting more than 3 months on the basis of clinical examination. Criteria for exclusion from the study will include: patients under 18 years of age, patients who are allergic to any ingredient of the preparation, pregnant or breast-feeding women, patients taking preparations that contain similar ingredients and/or have similar effects, obese patients, patients with active cancer, patients with severe systemic diseases, including genetic and neurological diseases, patients with severe mental illnesses, patients who are taking or in the last 12 months have taken antidepressants and/or myorelaxants and/or other drugs that affect neuromuscular activity, patients addicted to alcohol or drugs.

Qualified study participants will be randomly assigned to two groups. The studied group will receive an aqueous solution containing CBD and CBN, to drink at home in the dose determined by the attending physician, while the control group will receive an aqueous solution of placebo, to drink at home in the dose determined by the attending physician during this time. Each subject will be tested on the day of qualification (day 0), after 20 (day 20), and then 40 (day 40) and 60(day 60) days after the qualification day using the following methods:

* EMG (Electromyography) (day 0, day 20, day 40, day 60)
* Pressure pain threshold test (PPT) using the Wagner Paintest FPX 25 algometer (day 0, day 20, day 40, day 60)
* Clinical examination according to diagnostic criteria for temporomandibular disorders - DC / TMD International Examination Form (day 0, day 20, day 40, day 60)
* Surveys: Graded Chronic Pain Scale oraz McGill Pain Questionnaire (day 0, day 20, day 40, day 60), Satisfaction with Life Scale (day 0, day 20, day 40, day 60), Pittsburgh Sleep Quality Index (day 0, day 20, day 40, day 60), The Migraine Disability Assessment Test -MIDAS (day 0, day 20, day 40, day 60), Central Sensitisation Inventory (CSI) (day 0, day 20, day 40, day 60), Bruxscreen Q (day 0, day 20, day 40, day 60), Generalised Anxiety Disorder Assessment (day 0, day 20, day 40, day 60), Insomnia Severity Index (day 0, day 20, day 40, day 60), The Perceived Stress Scale (day 0, day 20, day 40, day 60), Somatic Symptom Scale - 8 (day 0, day 20, day 40, day 60)

ELIGIBILITY:
Inclusion Criteria:

* facial pain and headache of muscular origin for more than 3 months

Exclusion Criteria:

* patients under 18 years of age,
* patients who are allergic to any ingredient of the preparation,
* pregnant or breast-feeding women,
* patients taking preparations that contain similar ingredients and/or have similar effects,
* obese patients,
* patients with active cancer,
* patients with severe systemic diseases, including genetic and neurological diseases,
* patients with severe mental illnesses,
* patients who are taking or in the last 12 months have taken antidepressants and/or myorelaxants and/or other drugs that affect neuromuscular activity,
* patients addicted to alcohol or drugs.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2025-04-01 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
The influence of an aqueous solution containing CBD and CBN on muscle pain assessed using pressure pain threshold test (PPT) using the Wagner Paintest FPX 25 algometer. | 3 months
  Each participant will undergo pressure pain threshold test (PPT) using the Wagner Paintest FPX 25 algometer before and after taking an aqueous solution containing CBD and CBN.
The influence of an aqueous solution containing CBD and CBN on electrical activity and nerve conduction in muscles using EMG ( Electromyography). | 3 months
  Each participant will undergo EMG ( Electromyography) before and after taking an aqueous solution containing CBD and CBN. EMG measures the electrical activity of the muscle during rest, slight contraction and forceful contraction.

SECONDARY OUTCOMES:
The effectiveness of an aqueous solution containing CBD and CBN reduction on Facial Pain and Headache of Muscular Origin assessed by clinical examination in accordance to Diagnostic Criteria for Temporomandibular Disorders (DC/TMD) protocol. | 3 months
  Each patient will undergo DC/TMD protocol-based clinical examination before and after taking the aqueous solution containing CBD and CBN using DC/TMD examination form assessing incidence of pain of masticatory muscles and surrounding structures.
The influence of an aqueous solution containing CBD and CBN on reduction of Facial Pain and Headache of Muscular Origin using Pain Numerical Rating Scale. | 3 months
  Each participant will be asked to assess the pain during muscle palpation using Pain Numerical Rating Scale before and after taking the aqueous solution containing CBD and CBN. It is a subjective measure in which individuals rate their pain on an eleven-point numerical scale. The scale is composed of 0 (no pain at all) to 10 (worst imaginable pain).
The influence of an aqueous solution containing CBD and CBN on muscle pain assessed using Graded Chronic Pain Scale. | 3 months
  Each participant will fill in Graded Chronic Pain Scale. Scoring Criteria for Grading Chronic Pain Severity: Characteristic Pain Intensity is a 0 to 100 score derived from Questions 1 through 3:Mean (Pain Right Now, Worst Pain, Average Pain) X 10. Disability Score is 0 to 100score derived from Questions 4 through 6:Mean (Daily Activities, Social Activities, Work Activities) X 10. Disability Points: Add the indicated points for Disability Days (Question 7)and for Disability Score. Classification: GRADE 0- No TMD pain in prior 6 months. GRADE I-Low Intensity Characteristic Pain Intensity<50, Low Disability<3 Disability Point. GRADE II -High Intensity Characteristic Pain Intensity >50, LowDisability<3 Disability Points. GRADE III- High Disability3 to 4 Disability Points, Moderately Limiting (Regardless of Characteristic Pain Intensity). GRADE IV- High Disability 5 to 6 Disability Points, Severely Limiting (Regardless of Characteristic Pain Intensity).
The influence of an aqueous solution containing CBD and CBN on muscle pain assessed using McGill Pain Questionnaire. | 3 months
  Each participant will fill in McGill questionnaire that is composed of 78 words. Respondents choose those that best describe their experience of pain. Scores are tabulated by summing values associated with each word; scores range from 0 (no pain) to 78 (severe pain).
The influence of an aqueous solution containing CBD and CBN on muscle pain assessed using Pittsburgh Sleep Quality Index. | 3 months
  Each participant will fill in Pittsburgh Sleep Quality Index. The measure consists of 19 individual items, creating 7 components that produce one global score ranging from 0 to 21, where lower scores mean better sleep quality.
The influence of an aqueous solution containing CBD and CBN on muscle pain assessed using Satisfaction with Life Scale Questionnaire. | 3 months
  Each participant will fill in Satisfaction With Life Scale (SWLS). The SWLS is a 7-point Likert style response scale. The possible range of scores is 5-35, with a score of 20 representing a neutral point on the scale. Scores between 5-9 indicate the respondent is extremely dissatisfied with life, whereas scores between 31-35 indicate the respondent is extremely satisfied.
The influence of an aqueous solution containing CBD and CBN on muscle pain assessed using the Migraine Disability Assessment Test - MIDAS | 3 months
  The Migraine Disability Assessment Test (MIDAS) is a test used by doctors to determine how severely migraines affect a patient's life. Patients are asked questions about the frequency and duration of their headaches, as well as how often these headaches limited their ability to participate in activities at work, at school, or at home.
The influence of an aqueous solution containing CBD and CBN on muscle pain assessed by Central Sensitization Inventory | 3 months
  Each participant will fill in Central Sensitizatin Inventory. This questionnaire consist of two parts. First part includes 25 questions regarding common central sensitivity symptoms. It allows to categorize participant into one of five categories: subclinical (0-29), mild (30-39), moderate (40-49), severe (50-59), and extreme (60-100) Second part is not scored, but it determines if the participant has been diagnosed with certain CSS disorders or related disorders.
The influence of an aqueous solution containing CBD and CBN on muscle pain assessed by Bruxscreen Q questionnaire. | 3 months
  Each participant will fill in the Bruxscreen Q questionnaire which is a self-report outcome measure designed to identify patients who have symptoms that may be related to bruxism. There is 9 questions about clenching, grinding, jaw locking and other jaw symptoms, where frequent responding often or always indicates the possibility of having bruxism.
The influence of an aqueous solution containing CBD and CBN on muscle pain assessed by Generalized Anxiety Disorder -7 | 3 months
  Each participant will fill in Generalized Anxiety Disorder -7 that consists of 7 items. Total score ranges 0-21 points. Scores of 5, 10, and 15 are taken as the cut-off points for mild, moderate and severe anxiety, respectively.
The influence of an aqueous solution containing CBD and CBN on muscle pain assessed by Insomnia Severity Index (ISI) | 3 months
  Each participant will fill in Insomnia Severity Scale. Questionnaire contains 5 questions, scored from 0 to 4 depending on the severity of ailments. Minimal score is 0, maximal score is 20. A total point value of up to 10 is considered the norm, while a score above 14 points indicates clinically significant insomnia.
The influence of an aqueous solution containing CBD and CBN on muscle pain assessed by Perceived Stress Scale -10 | 3 months
  Each participant will fill in Perceived Stress Scale -10. Scores are obtained by reversing the scores on the four positive items, e.g., 0=4, 1=3, 2=2, etc. and then summing across all 10 items. Items 4,5, 7, and 8 are the positively stated items. It can range from 0 to 40. Scores ranging from 0-13 would be considered low stress,14-26 would be considered moderate stress, 27-40 would be considered high perceived stress.
The influence of an aqueous solution containing CBD and CBN on muscle pain assessed by Somatic Symptom Scale - 8 | 3 months
  Each participant will fill in the Somatic Symptom Scale - 8 (SSS-8) which is a brief self-report questionnaire used to assess somatic symptom burden. It measures the perceived burden of common somatic symptoms. These symptoms were originally chosen to reflect common symptoms in primary care but they are relevant for a large number of diseases and mental disorders. Scoring: 0-3: no to minimal, 4-7: low, 8-11: medium,12-15: high,16-32: very high.

CONTACTS AND LOCATIONS:
Locations (1):
- Wroclaw Medical University, Wroclaw, Poland

IPD SHARING:
Plan to Share IPD: No